CLINICAL TRIAL: NCT00748475
Title: Countering Stimulus-Induced Alpha-Desynchronization to Treat Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Nathan Weisz, Dr. Nathan Weisz, University of Konstanz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TE0602-1
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurofeedback (Experimental)
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback

SUMMARY:
The purpose of the study is to examine the effect of alpha-neurofeedback while subjects listen to a noise on tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Duration of Tinnitus >= 6 months and <= 20 years
* Subjective Tinnitus

Exclusion Criteria:

* History of neurological or more than mild psychiatric diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Reduction of tinnitus distress using the Tinnitus Questionaire | Before the first and after the last session.
Cortical Alpha Power | Before the first and after the last session

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Weisz, PhD, Principal Investigator — University Konstanz; Thomas Hartmann, Dipl.-Psych., Study Chair — University Konstanz